CLINICAL TRIAL: NCT00465101
Title: A Prospective Clinical Study for GreenLight HPS in the Treatment of Obstructive Benign Prostatic Hyperplasia (BPH)
Brief Title: A Long-Term Study Examining the Treatment of Benign Prostatic Hyperplasia With Photoselective Vaporization
Acronym: PVP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PE0603
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Results first posted 2015-10-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2012-06

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; Transurethral resection of the prostate; Lower urinary tract symptoms; GreenLight; Laserscope; Photoselective vaporization of the prostate; enlarged prostate
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GreenLight HPS (Other)
  Interventions: Device: GreenLight HPS

INTERVENTIONS:
Device: GreenLight HPS — Greenlight HPS laser system for treatment of BPH

SUMMARY:
To gain clinical experience with the GreenLight HPS System, a system designed to vaporize and coagulate tissue in the treatment of benign prostatic hyperplasia to reduce lower urinary tract symptoms.

DETAILED DESCRIPTION:
Enlarged prostate or Benign Prostatic Hyperplasia (BPH) is one of the most common diseases of aging men and can be associated with lower urinary tract symptoms (LUTS) such as having to urinate very often, a sudden strong feeling of having to urinate, having to get up at night to urinate, decreased and intermittent force of stream and the feeling of incomplete bladder emptying. These symptoms affect quality of life by interfering with normal daily activities and sleep patterns. When surgery is the best treatment option for the patient, the most common technique is a "transurethral resection of the prostate" (TURP). TURP involves removing the some of the extra tissue of the prostate gland. Even though TURP is a good treatment, there are concerns about the frequency of complications following treatment as well as the significant costs to patients, doctors, and insurance providers.

Photoselective vaporization of the prostate (PVP) is a relatively new technology that has similar benefits with fewer side effects than TURP. PVP is a minimally invasive procedure that uses a special high-energy laser to eliminate excess prostate tissue and seal the treated area. This technology has been used for more than a decade with over 200,000 procedures performed worldwide.

The focus of this study is to 1) document the long-term advantages of GreenLight HPS 120w and 2) to show that the stronger laser is a more flexible and efficient device which allows for a shorter procedure time, may be done in an out-patient setting in healthy patients, allows for shorter catheterization time, may result in a rapid urinary flow rate with minimal side effects, and may allow a quick return to normal activities. This device has been approved by the United States Food and Drug Administration (FDA) for treatment of obstructive BPH.

ELIGIBILITY:
Inclusion Criteria:

* All male subjects ≥ 45 years of age who have a history of symptomatic/obstructive symptoms secondary to BPH greater than 3 months, an International Prostate Symptom Score (IPSS) / American Urology Association (AUA) score >14, require surgical intervention, and are an acceptable risk for anesthesia and surgery are eligible to participate in this study

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) classification of physical status > III
* An unstable cardiopulmonary disorder, previously or recently diagnosed by standard methods
* A myocardial infarction or coronary artery stent placement within 6 months of the treatment
* Neurogenic lower urinary dysfunction
* A post-void residual (PVR) volume ≥ 400 mL
* Pre-existing urinary incontinence
* Active localized or systemic infection, including urinary tract infection (UTI) or prostatitis affecting bladder function
* Pre-existing damage of external urinary sphincter
* Presence of cystolithiasis, urethral stricture, or bladder neck contracture
* Prostate volume (PV), as measured by transrectal ultrasound (TRUS), less than 30cc or greater than 200cc
* Previously confirmed or suspected malignancy of prostate or bladder, treated or untreated
* Immunocompromised subjects
* Serious bleeding disorders and coagulopathy. For example: hemophilia or Von Willebrand's disease
* Desire to preserve antegrade ejaculation
* Calcification of prostate tissue, usually after severe prostatitis
* Deemed unfit for laser vaporization as determined by the attending physician
* Enrollment in a concurrent clinical trial of any treatment (drug or device) that could affect urogenital function without sponsors' approval
* Unable or unwilling to sign the Informed Consent Form (ICF) and/or comply with all follow-up requirements

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-05; Primary Completion 2012-08 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claus G Roehrborn, MD, Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (9):
- United States (9):
  - UCLA, Los Angeles, California
  - Connecticut Clinical Reseach Center, Middlebury, Connecticut
  - North Fulton Urology, P.C., Roswell, Georgia
  - Affiliates in Urology, Detroit, Michigan
  - PC Group/Universtiy Urology Association, New York, New York
  - Glickman Urological Institute, Cleveland, Ohio
  - Oklahoma University Health Science Center_Urology, Oklahoma City, Oklahoma
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Urology of Virginia, Virginia Beach, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients at least 45 years of age with symptomatic/obstructive BPH for at least 3 months and requiring surgical intervention. Enrollment occurred at 10 academic and private medical centers in the US. The last patient follow up visit was completed in August 2012. The last site close-out visit was completed January 2013.
Groups:
- GreenLight HPS Laser System: GreenLight HPS Laser System therapy for patients with BPH.
Period: Overall Study
Arm/Group | GreenLight HPS Laser System
Started | 150
Completed | 91
Not Completed | 59
Not completed — Aborted Proc./Treatment Not Attempted | 3
Not completed — Change in health precluded follow up | 4
Not completed — Did not meet study criteria | 4
Not completed — Lost to Follow-up | 5
Not completed — Other | 6
Not completed — Pt. Insurance not accepted at center | 2
Not completed — Patient postponed procedure | 1
Not completed — Site closed due to IRB expiration | 1
Not completed — Unable to obtain IRB approval | 1
Not completed — Death | 3
Not completed — Withdrawal by Subject | 25
Not completed — Physician Decision | 1
Not completed — Withdrew consent prior to procedure | 3

BASELINE CHARACTERISTICS:
Arm/Group | GreenLight HPS Laser System
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 150
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 148
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 150
Height (cm) [Mean (Standard Deviation); unit: cm] | 178.5 (7.0)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 87.3 (14.8)
Smoker [Number; unit: participants] | 10
Previous BPH Treatment [Number; unit: participants] | 134
Average Duration of Obstructive Symptoms (months) [Mean (Standard Deviation); unit: months] | 74.9 (60.2)
Peak Flow Rate (ml/sec) [Mean (Standard Deviation); unit: ml/sec] | 10.7 (5.4)
Post-void Residual Volume (ml) [Mean (Standard Deviation); unit: ml] | 112.5 (115.5)
Serum Prostate Specific Antigen (PSA) level (ng/ml) [Mean (Standard Deviation); unit: ng/ml] | 2.5 (2.1)
Prostate Volume (cc) [Mean (Standard Deviation); unit: cc] | 58.5 (28.4)
International Prostate Symptom Score (IPSS) at Baseline [Mean (Standard Deviation); unit: Scores on a scale] — The IPSS measures the severity of BPH symptoms and is calculated as the sum of 7-items from a participant-administered instrument. The IPSS ranges from 0 (asymptomatic) to 35 (severely symptomatic) with higher values indicating a worse condition.
  Scores on a scale | 22.9 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Success
Description: Treatment success is determined on a per patient basis and is defined as [(baseline I-PSS - I-PSS at 6-months)/ baseline I-PSS] greater than or equal to 50%
Time Frame: 6 months
Population: Participants who received the study treatment and for whom the outcome measure is available.
Measure: Number; unit: percentage of participants
Arm/Group | GreenLight HPS Laser System
Number analyzed (Participants) | 119
percentage of participants | 84.9

2. Secondary Outcome: Treatment-related Complication
Description: Treatment-related events include the following:
  * Infection that requires IV antibiotics or re-hospitalization or prolongation of existing hospitalization
  * Perforation / injury of adjacent organ(s)
  * Bladder neck contracture(s) requiring re-catheterization after post-surgery catheter removal
  * Hematuria requiring transfusion
  * Urinary retention requiring corrective intervention
  * De novo erectile dysfuction (ED)
  * Transfusion secondary to procedure-related anemia
  * Post procedure incontinence secondary to damage to the external urinary sphincter
  * Any other treatment-related injury requiring intervention
Time Frame: 3 months
Population: Participants who received the study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of subjects with complication
Arm/Group | Treatment Related Complication at 3 Months
Number analyzed (Participants) | 135
percentage of subjects with complication | 11.1 [6.5 to 17.0]

3. Secondary Outcome: Percentage of Participants With Clinically-significant Improvement in Uroflow.
Description: A clinically significant improvement in uroflow is defined as an increase in peak urinary flow rate (Qmax) of at least five ml/sec from baseline to 6 months
Time Frame: 6 months post-treatment
Population: Participants who received the study treatment and for whom the outcome measure is available.
Measure: Number (95% Confidence Interval); unit: percentage of patients improved
Groups:
- Number of Subjects With Baseline and 6 Month Values: The total number of patients that treated equals 136; the total number of patients with Baseline and 6 month values equals 117.
Arm/Group | Number of Subjects With Baseline and 6 Month Values
Number analyzed (Participants) | 117
percentage of patients improved | 70.9 [61.8 to 79.0]

4. Secondary Outcome: Percentage of Participants With Clinically-significant Improvement in Post-void Residual Urine Volume.
Description: A clinically significant improvement in post-void residual is defined as a decrease of at least 50ml from baseline to 6 months.
Time Frame: 6 months post-treatment
Population: Participants who received the study treatment and for whom the outcome measure is available.
Measure: Number (95% Confidence Interval); unit: percentage of patients improved
Arm/Group | Number of Subjects With Baseline and 6 Month Values
Number analyzed (Participants) | 117
percentage of patients improved | 42.7 [33.6 to 52.2]

5. Secondary Outcome: Quality of Life Score (QoL) From I-PSS From Baseline Through 5 Years.
Description: Participant response to the question "If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that?". Values range from 0 ("Delighted") to 6 ("Terrible") with higher values indicating worse outcomes.
Time Frame: 5 years
Population: Participants who received the study treatment and for whom the outcome measure is available.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Baseline QoL Score | 3 Months | 6 Months | 1 Year | 2 Years | 3 Years | 4 Years | 5 Years
Number analyzed (Participants) | 136 | 131 | 119 | 117 | 103 | 97 | 59 | 4
Score on a scale | 4.4 (1.1) | 1.6 (1.4) | 1.3 (1.2) | 1.3 (1.2) | 1.3 (1.2) | 1.3 (1.3) | 1.2 (1.2) | 0.8 (1.0)

6. Secondary Outcome: Gross Hematuria
Description: Kaplan-Meier estimate of percentage of participants who require a blood transfusion as a result of hematuria.
Time Frame: 91 days
Population: Participants who received the study treatment
Measure: Number; unit: Percentage of subjects
Arm/Group | Peri-Operative (0-14 Days) | Delayed (15-91 Days)
Number analyzed (Participants) | 136 | 136
Percentage of subjects | 1.5 | 2.2

7. Secondary Outcome: Percentage of Participants With Treatment Success
Description: Treatment success is determined on a per patient basis and is defined as a 50% or greater decrease in IPSS from baseline to the specified time point.
Time Frame: 5 Years
Population: Participants who received the study treatment and for whom the outcome measure is available.
Measure: Number (95% Confidence Interval); unit: Percent of subjects w/ treatment success
Arm/Group | Baseline | 3 Months | 6 Months | 1 Year | 2 Years | 3 Year | 4 Years | 5 Years
Number analyzed (Participants) | 136 | 131 | 119 | 117 | 103 | 97 | 59 | 4
Percent of subjects w/ treatment success | 0 [0 to 0] | 72.5 [64.0 to 80.0] | 84.9 [77.2 to 90.8] | 77.8 [69.2 to 84.9] | 79.6 [70.5 to 86.9] | 75.3 [65.5 to 83.5] | 74.6 [61.6 to 85.0] | 100.0 [39.8 to 100.0]

8. Secondary Outcome: Length of Time to Return to Pre-treatment Level of Physical Activity (in Days), Excluding Sexual Activity.
Time Frame: Up to five years
Population: Participants who received the study treatment and for whom the outcome measure is available.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Return to Activity (Days)
Number analyzed (Participants) | 126
days | 9.5 (9.6)

9. Other Pre Specified Outcome: Length of Hospital Stay (LOS)
Description: Defined as the time from admission to the healthcare facility until discharge (in hours).
Time Frame: Peri-Operative Period
Population: Participants who received the study treatment and for whom the outcome measure is available.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Length of Hospital Stay (Hours)
Number analyzed (Participants) | 135
hours | 5.2 (7.1)

10. Other Pre Specified Outcome: Length of Catheterization (LOC)
Description: Defined as the time the subject required an indwelling Foley catheter post treatment (in hours).
Time Frame: Recovery Period
Population: Participants who received the study treatment and for whom the outcome measure is available.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Length of Catheterization
Number analyzed (Participants) | 124
hours | 21.9 (22.9)

11. Other Pre Specified Outcome: Length of Procedure (LOP)
Description: Defined as the time from cystoscope insertion into the urethra to the time of cystoscope removal (in minutes).
Time Frame: Procedure
Population: Participants who received the study treatment and for whom the outcome measure is available.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Length of Procedure (Min)
Number analyzed (Participants) | 136
minutes | 53.9 (21.5)

12. Other Pre Specified Outcome: Length of Lasing (LOL)
Description: Total time the laser was on during the study procedure.
Time Frame: Procedure
Population: Participants who received the study treatment and for whom the outcome measure is available.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Length of Lasing Time
Number analyzed (Participants) | 135
minutes | 34.1 (17.5)

13. Other Pre Specified Outcome: Number of Fibers Used During Procedure
Time Frame: Procedure
Population: Participants who received the study treatment and for whom the outcome is available.
Measure: Mean (Standard Deviation); unit: number of fibers used
Arm/Group | Number of Fibers Used
Number analyzed (Participants) | 136
number of fibers used | 1.2 (0.5)

14. Other Pre Specified Outcome: Total Joules Used
Description: Total energy applied during the study procedure
Time Frame: Procedure
Population: Participants who received the study treatment and for whom the outcome measure is available.
Measure: Mean (Standard Deviation); unit: kilojoules (kJ)
Arm/Group | Total Energy Delivered
Number analyzed (Participants) | 135
kilojoules (kJ) | 190.6 (94.4)

15. Secondary Outcome: Occurrence of Retrograde Ejaculation
Description: Kaplan-Meier estimate of percentage of participants who experience retrograde ejaculation.
Time Frame: 5 Year Follow Up
Population: Participants who received the study treatment
Measure: Number (95% Confidence Interval); unit: percentage of subjects with RE
Arm/Group | Retrograde Ejaculation Occurrence Rate
Number analyzed (Participants) | 136
percentage of subjects with RE | 43.3 [34.1 to 52.0]

ADVERSE EVENTS:
Time Frame: Through study completion; planned to be 5 years.
Description: All participants who received the study treatment will be considered at risk of having an adverse event. This study allowed adverse events to be collected not using specific event terms (e.g., "Other" adverse events).
Arm/Group | GreenLight HPS Laser System
Serious Adverse Events (participants affected / at risk) | 35/136
Other Adverse Events (participants affected / at risk) | 97/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GreenLight HPS Laser System (N=136)
Allergic Reaction / Hypersensitivity (General disorders) | 1 (1)
Infection (other than UTI) (Infections and infestations) | 1 (1)
Perforation - Prostate (Renal and urinary disorders) | 2 (2)
Injury - Other (General disorders) | 1 (1)
Pain / Discomfort - Leg (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain / Discomfort - Other (General disorders) | 4 (4)
Bladder Neck Contracture / Outlet Obstruct (Renal and urinary disorders) | 1 (1)
Hematuria - Gross (Renal and urinary disorders) | 1 (2)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Deep Venous Thrombosis (Vascular disorders) | 1 (1)
Other: Death (General disorders) | 2 (2)
Other: Prostate Cancer (Renal and urinary disorders) | 3 (3)
Other: Renal Failure - Acute (Renal and urinary disorders) | 1 (1)
Other: Atrial Arrhythmia (Cardiac disorders) | 2 (2)
Other: Hernia (Musculoskeletal and connective tissue disorders) | 1 (1)
Other: Lymphoma (Blood and lymphatic system disorders) | 1 (1)
Other: Cardiomyopathy (Cardiac disorders) | 1 (1)
Other: Coronary Artery Disease (Vascular disorders) | 2 (3)
Other: Multiple Myeloma (Musculoskeletal and connective tissue disorders) | 1 (1)
Other: Rotator Cuff Tear (Musculoskeletal and connective tissue disorders) | 2 (2)
Other: Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other: Epistaxis (Blood and lymphatic system disorders) | 1 (1)
Other: Stroke (Vascular disorders) | 2 (2)
Other: Knee Replacement (Musculoskeletal and connective tissue disorders) | 1 (1)
Other: Obesity - Worsening (Metabolism and nutrition disorders) | 1 (1)
Other (General disorders) | 5 (8)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GreenLight HPS Laser System (N=136)
Dysuria (Renal and urinary disorders) | 30 (31)
Retrograde Ejaculation - De Novo (Renal and urinary disorders) | 30 (30)
Urinary Urgency (Renal and urinary disorders) | 24 (24)
Retrograde Ejaculation (Renal and urinary disorders) | 23 (23)
Urinary Frequency (Renal and urinary disorders) | 14 (15)
Urinary Tract Infection (UTI) (Renal and urinary disorders) | 9 (9)
Hematuria (Renal and urinary disorders) | 15 (15)
Hematuria - Gross (Renal and urinary disorders) | 9 (10)
Erectile Dysfunction - De Novo (Renal and urinary disorders) | 8 (8)
Urinary Incontinence - De Novo (Renal and urinary disorders) | 10 (10)
Pain / Discomfort - Other (General disorders) | 6 (6)
Allergic Reaction / Hypersensitivity Reaction (General disorders) | 1 (1)
Bladder Neck Contracture / Outlet Obstruct (Renal and urinary disorders) | 4 (6)
Prostatitis (Renal and urinary disorders) | 5 (5)
Urinary Retention - Acute (Renal and urinary disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 2 (2)
Erectile Dysfunction - Worsening (Renal and urinary disorders) | 1 (1)
Perforation - Prostate (Renal and urinary disorders) | 2 (2)
Sloughing (Renal and urinary disorders) | 1 (1)
Urethral Stricture (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Other: Nocturia (Renal and urinary disorders) | 4 (4)
Other: Urinary Dribbling (Renal and urinary disorders) | 6 (7)
Other: Hypertension (Cardiac disorders) | 1 (1)
Other: Bladder Spasm (Renal and urinary disorders) | 3 (3)
Other: Lack of Sensation During Ejaculation (Renal and urinary disorders) | 2 (2)
Other: Overactive Bladder (Renal and urinary disorders) | 2 (2)
Other: Paraphimosis (Skin and subcutaneous tissue disorders) | 1 (1)
Other: Urethral Burning at Foley Catheter Site (Renal and urinary disorders) | 2 (2)
Other: Urine Flow Decreased Force (Renal and urinary disorders) | 1 (1)
Other: Bladder Pressure (Renal and urinary disorders) | 1 (1)
Other: Clot Retention (Renal and urinary disorders) | 1 (1)
Other: Decrease Sense of Emptying Bladder (Renal and urinary disorders) | 1 (1)
Other: Sexual Dysfunction (Reproductive system and breast disorders) | 1 (1)
Other (General disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Follow-up of subjects was discontinued in August 2012 prior to most participants completing the assessment planned at 5 years. At the time of the discontinuation, all but five of the participants remaining on study had completed 3 years of follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No